CLINICAL TRIAL: NCT03353350
Title: A 56-week, Multicenter, Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of Efpeglenatide Once Weekly in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Diet and Exercise
Brief Title: Efficacy and Safety of Efpeglenatide Versus Placebo in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Diet and Exercise
Acronym: AMPLITUDE-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14822; 2016-001857-42; U1111-1182-1806 (Other: UTN)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — efpeglenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Efpeglenatide 2mg (Experimental): Efpeglenatide low dose (Prefilled syringe) administered once weekly for 56 weeks
  Interventions: Drug: efpeglenatide (SAR439977)
- Efpeglenatide 4 mg (Experimental): Efpeglenatide middle dose (Prefilled syringe) administered once weekly for 56 weeks (including titration period)
  Interventions: Drug: efpeglenatide (SAR439977)
- Efpeglenatide 6 mg (Experimental): Efpeglenatide high dose (Prefilled syringe) administered once weekly for 56 weeks (including titration period)
  Interventions: Drug: efpeglenatide (SAR439977)
- Placebo (Placebo Comparator): Matching placebo (Prefilled syringe) administered once weekly for 56 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: efpeglenatide (SAR439977) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: Efpeglenatide 2mg; Efpeglenatide 4 mg; Efpeglenatide 6 mg
Drug: placebo — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo in glycated hemoglobin (HbA1c) change in participants with T2DM (Type 2 Diabetes Mellitus) inadequately controlled with diet and exercise.

Secondary Objectives:

* To demonstrate the superiority of once-weekly injection of efpeglenatide in comparison to placebo on glycemic control
* To demonstrate the superiority of once-weekly injection of efpeglenatide in comparison to placebo on body weight
* To evaluate the safety of once-weekly injection of efpeglenatide

DETAILED DESCRIPTION:
Study duration per participant is approximately 65 weeks, including a 3-week screening period, 30 weeks core treatment period, 26 weeks extension treatment period, and 6 weeks safety follow up.

ELIGIBILITY:
Inclusion criteria:

* Participants must be at least 18 years of age at the time of signing the informed consent.
* Participants with T2DM, and treated with diet and exercise.
* Hemoglobin A1c between 7.0% and 10.0% (inclusive) measured by the central laboratory at Screening.

Exclusion criteria:

* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to) gastroparesis, unstable and not controlled gastroesophageal reflux disease within 6 months prior to Screening or history of surgery affecting gastric emptying.
* History of pancreatitis (unless pancreatitis was related to gallstone and cholecystectomy has been performed) and pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, and pancreatectomy.
* Personal or family history of Medullary Thyroidian Cancer (MTC) or genetic conditions that predisposes to MTC (eg multiple endocrine neoplasia syndromes).
* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months of screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Body weight change of ≥5 kg within the last 3 months prior to Screening.
* Systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg at Randomization.
* End-stage renal disease as defined by estimated glomerular filtration rate (eGFR , by Modification of Diet in Renal Disease [MDRD]) of <15 mL/min/1.73 m2.
* Laboratory findings at the Screening Visit:
* Alanine aminotransferase (ALT ) or aspartate aminotransferase (AST ) >3 times the upper limit of the normal (ULN ) or total bilirubin >1.5 times the ULN (except in case of documented Gilbert's syndrome).
* Amylase and/or lipase: >3 times the ULN laboratory range.
* Calcitonin ≥5.9 pmol/L (20 pg/mL).
* Gastric surgery or other gastric procedures intended for weight loss within 2 years prior to Screening, or planned during study period.
* History of drug or alcohol abuse within 6 months prior to the time of Screening.
* Pregnant (demonstrated by serum pregnancy test at Screening) or breast-feeding women.
* Women of childbearing potential not willing to use highly effective method(s) of birth control during the study period and for at least 5 weeks after the last dose of study intervention.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (54):
- United States (32):
  - Investigational Site Number 8400004, Birmingham, Alabama
  - Investigational Site Number 8400005, Glendale, Arizona
  - Investigational Site Number 8400003, Canoga Park, California
  - Investigational Site Number 8400007, Chula Vista, California
  - Investigational Site Number 8400011, La Mesa, California
  - Investigational Site Number 8400009, Los Angeles, California
  - Investigational Site Number 8400029, Pomona, California
  - Investigational Site Number 8400024, Tarzana, California
  - Investigational Site Number 8400026, Van Nuys, California
  - Investigational Site Number 8400010, DeLand, Florida
  - Investigational Site Number 8400006, Hialeah, Florida
  - Investigational Site Number 8400032, West Palm Beach, Florida
  - Investigational Site Number 8400025, Lawrenceville, Georgia
  - Investigational Site Number 8400034, Chicago, Illinois
  - Investigational Site Number 8400033, Kansas City, Missouri
  - Investigational Site Number 8400018, Lincoln, Nebraska
  - Investigational Site Number 8400062, Las Vegas, Nevada
  - Investigational Site Number 8400021, Las Vegas, Nevada
  - Investigational Site Number 8400001, Bridgeton, New Jersey
  - Investigational Site Number 8400028, Burlington, North Carolina
  - Investigational Site Number 8400031, Wilmington, North Carolina
  - Investigational Site Number 8400013, Maumee, Ohio
  - Investigational Site Number 8400008, Hatboro, Pennsylvania
  - Investigational Site Number 8400017, Carrollton, Texas
  - Investigational Site Number 8400030, Dallas, Texas
  - Investigational Site Number 8400015, Houston, Texas
  - Investigational Site Number 8400019, Plano, Texas
  - Investigational Site Number 8400020, San Antonio, Texas
  - Investigational Site Number 8400016, San Antonio, Texas
  - Investigational Site Number 8400027, San Antonio, Texas
  - Investigational Site Number 8400023, Schertz, Texas
  - Investigational Site Number 8400002, Holladay, Utah
- Germany (3):
  - Investigational Site Number 2760005, Berlin
  - Investigational Site Number 2760003, Frankfurt am Main
  - Investigational Site Number 2760001, Leipzig
- Poland (7):
  - Investigational Site Number 6160005, Gdansk
  - Investigational Site Number 6160004, Gdynia
  - Investigational Site Number 6160007, Katowice
  - Investigational Site Number 6160002, Krakow
  - Investigational Site Number 6160006, Poznan
  - Investigational Site Number 6160003, Warsaw
  - Investigational Site Number 6160001, Wroclaw
- Ukraine (4):
  - Investigational Site Number 8040003, Kyiv
  - Investigational Site Number 8040001, Kyiv
  - Investigational Site Number 8040002, Kyiv
  - Investigational Site Number 8040004, Vinnitsa
- United Kingdom (8):
  - Investigational Site Number 8260005, Birmingham
  - Investigational Site Number 8260004, Cardiff
  - Investigational Site Number 8260007, Chorley
  - Investigational Site Number 8260008, Glasgow
  - Investigational Site Number 8260001, Hexham
  - Investigational Site Number 8260003, Liverpool
  - Investigational Site Number 8260006, Manchester
  - Investigational Site Number 8260002, Reading

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frias JP, Choi J, Rosenstock J, Popescu L, Niemoeller E, Muehlen-Bartmer I, Baek S. Efficacy and Safety of Once-Weekly Efpeglenatide Monotherapy Versus Placebo in Type 2 Diabetes: The AMPLITUDE-M Randomized Controlled Trial. Diabetes Care. 2022 Jul 7;45(7):1592-1600. doi: 10.2337/dc21-2656. PMID 35671039

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo (Prefilled syringe) administered once weekly for 56 weeks
  placebo: Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
- Efpeglenatide 2 mg: Efpeglenatide low dose (Prefilled syringe) administered once weekly for 56 weeks
  efpeglenatide (SAR439977): Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
- Efpeglenatide 4 mg: Efpeglenatide middle dose (Prefilled syringe) administered once weekly for 56 weeks (including titration period)
  efpeglenatide (SAR439977): Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
- Efpeglenatide 6 mg: Efpeglenatide high dose (Prefilled syringe) administered once weekly for 56 weeks (including titration period)
  efpeglenatide (SAR439977): Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
Period: 30-week Core Treatment Period
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Started | 102 | 100 | 101 | 103
Completed | 80 | 81 | 77 | 81
Not Completed | 22 | 19 | 24 | 22
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Other: Not related to COVID-19 | 2 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 19 | 12 | 19 | 19
Period: 26-week Treatment Extension Period
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Started | 80 | 81 | 77 | 81
Completed | 75 | 78 | 73 | 67
Not Completed | 5 | 3 | 4 | 14
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Other: Not related to COVID-19 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Total
Number analyzed (Participants) | 102 | 100 | 101 | 103 | 406
Age, Customized [Count of Participants; unit: Participants] — Age group (years)
  Participants
    <50 | 22 | 21 | 30 | 21 | 94
    ≥50 and <65 | 43 | 46 | 44 | 44 | 177
    ≥65 and <75 | 26 | 28 | 20 | 31 | 105
    ≥75 | 11 | 5 | 7 | 7 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 45 | 49 | 42 | 187
  Male | 51 | 55 | 52 | 61 | 219
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 90 | 93 | 86 | 92 | 361
  Race : Black or African American | 10 | 6 | 13 | 8 | 37
  Race : Asian | 2 | 0 | 1 | 2 | 5
  Race : Other | 0 | 0 | 1 | 1 | 2
  Race : Multiple | 0 | 1 | 0 | 0 | 1
  Ethnicity : Hispanic or Latino | 20 | 20 | 25 | 21 | 86
  Ethnicity : Not Hispanic or Latino | 82 | 80 | 76 | 82 | 320
Region of Enrollment [Number; unit: participants]
  North America | 54 | 53 | 57 | 58 | 222
  Europe | 48 | 47 | 44 | 45 | 184
Screening HbA1c [Mean (Standard Deviation); unit: %] | 7.98 (0.85) | 8.03 (0.75) | 8.14 (0.93) | 8.07 (0.91) | 8.05 (0.87)
Baseline BMI [Mean (Standard Deviation); unit: kg/m²] | 34.8 (7.1) | 34.4 (6.4) | 33.8 (6.6) | 33.8 (6.9) | 34.2 (6.8)
Baseline BMI category [Count of Participants; unit: Participants]
  <30 | 28 | 28 | 28 | 28 | 112
  ≥30 and <40 | 52 | 53 | 58 | 60 | 223
  ≥40 | 22 | 19 | 15 | 14 | 70
  Unknown | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) (%)
Description: Change from Baseline to Week 30 in HbA1c
Time Frame: Baseline to Week 30
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
HbA1c (%) | -0.46 (1.16) | -1.14 (0.96) | -1.48 (1.01) | -1.59 (1.04)

2. Secondary Outcome: Change in HbA1c (%)
Description: Change from Baseline to Week 56 in HbA1c
Time Frame: Baseline to Week 56
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
HbA1c (%) | -0.52 (1.18) | -1.18 (0.79) | -1.51 (0.99) | -1.51 (0.18)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from Baseline to Week 30 in FPG
Time Frame: Baseline to Week 30
Measure: Mean (Standard Deviation); unit: FPG (mmol/L)
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
FPG (mmol/L) | 8.59 (2.13) | -0.87 (3.27) | 6.84 (1.57) | 6.55 (1.30)

4. Secondary Outcome: HbA1c <7%
Description: Number of participants with HbA1c <7.0% at Week 30
Time Frame: Week 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
Participants | 26 | 60 | 66 | 76

5. Secondary Outcome: Change in Body Weight at Week 30
Description: Change from Baseline to Week 30 in body weight
Time Frame: Baseline to Week 30
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
kg | -1.35 (3.15) | -1.01 (3.66) | -3.34 (4.19) | -3.19 (4.77)

6. Secondary Outcome: Change in Body Weight at Week 56
Description: Change from Baseline to Week 56 in body weight
Time Frame: Baseline to Week 56
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 100 | 101 | 103
kg | -1.26 (4.19) | -0.94 (4.96) | -3.24 (6.42) | -1.82 (5.52)

7. Secondary Outcome: Hypoglycemic Participants
Description: Number of participants with at least 1 hypoglycemic event during treatment period
Time Frame: Baseline to Week 56
Population: Safety population: All participants randomly assigned to IMP and who take at least 1 dose of IMP. Participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 102 | 103 | 99
Participants | 2 | 10 | 14 | 14

8. Secondary Outcome: Hypoglycemic Events
Description: Number of hypoglycemic events
Time Frame: Baseline to Week 56
Population: as for outcome 7
Measure: Number; unit: Number of events
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 102 | 103 | 99
Number of events | 2 | 10 | 14 | 14

9. Secondary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs
Time Frame: Baseline to Week 56
Population: as for outcome 7
Measure: Number; unit: Number of Treatment Emergent AEs
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 102 | 102 | 103 | 99
Number of Treatment Emergent AEs | 79 | 80 | 79 | 83

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs), Serious AEs (SAEs), Adverse Events of Special Interest (AESIs) and AEs requiring specific monitoring were collected from the date of signing the Informed Consent Form (ICF) until the end of the study, defined by the protocol for that participant as Week 62.
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102 | 0/103 | 1/99
Serious Adverse Events (participants affected / at risk) | 9/102 | 11/102 | 6/103 | 6/99
Other Adverse Events (participants affected / at risk) | 70/102 | 69/102 | 73/103 | 77/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Efpeglenatide 2 mg (N=102) | Efpeglenatide 4 mg (N=103) | Efpeglenatide 6 mg (N=99)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | Efpeglenatide 2 mg (N=102) | Efpeglenatide 4 mg (N=103) | Efpeglenatide 6 mg (N=99)
Nasopharyngitis (Infections and infestations) | 8 | 10 | 7 | 11
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 5 | 6
Viral upper respiratory tract infection (Infections and infestations) | 7 | 3 | 5 | 6
Bronchitis (Infections and infestations) | 4 | 3 | 3 | 4
Cystitis (Infections and infestations) | 3 | 2 | 1 | 1
Influenza (Infections and infestations) | 3 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 6 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 2 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 1
Otitis externa (Infections and infestations) | 1 | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 1
Body tinea (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 0
Ear infection (Infections and infestations) | 3 | 1 | 2 | 0
Eyelid infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tonsilitis (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadentis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 2 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 11 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 2
Stress (Psychiatric disorders) | 2 | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 6 | 10 | 15
Dizziness (Nervous system disorders) | 6 | 2 | 10 | 6
Paraesthesia (Nervous system disorders) | 2 | 1 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 2
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 3
Cataract (Eye disorders) | 1 | 1 | 1 | 2
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 2
Astigmatism (Eye disorders) | 0 | 1 | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Eyelid cyst (Eye disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0 | 0
Hypoaesthesia eye (Eye disorders) | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0 | 0
Presbyopia (Eye disorders) | 0 | 1 | 0 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 2 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertico (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 3
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 4 | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 2 | 4 | 2
Angina pectoris (Cardiac disorders) | 2 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular septal defect acquired (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 8 | 3 | 6
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 2 | 0 | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 9 | 17 | 25
Nausea (Gastrointestinal disorders) | 2 | 6 | 15 | 22
Constipation (Gastrointestinal disorders) | 6 | 9 | 14 | 16
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 7 | 12
Vomiting (Gastrointestinal disorders) | 0 | 3 | 8 | 9
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 5 | 8
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2 | 7
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 2 | 2
Eructation (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic steatosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 4 | 2 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2 | 2
Athralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ankle impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 3 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Mixed incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 6 | 9 | 11 | 11
Fatigue (General disorders) | 3 | 3 | 4 | 5
Injection site bruising (General disorders) | 3 | 3 | 2 | 3
Asthenia (General disorders) | 1 | 1 | 3 | 2
Chest pain (General disorders) | 2 | 1 | 3 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Injection site discomfort (General disorders) | 0 | 0 | 2 | 1
Injection site haemorrhage (General disorders) | 2 | 0 | 0 | 1
Injection site inflammation (General disorders) | 0 | 0 | 0 | 1
Injection site mass (General disorders) | 0 | 0 | 0 | 1
Injection site paraesthesia (General disorders) | 1 | 1 | 0 | 1
Injection site pruritus (General disorders) | 1 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Drug intolerance (General disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 1 | 0
Injection site vesicles (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 0
Medical device site reaction (General disorders) | 0 | 1 | 0 | 0
Medical device site vesicles (General disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 8 | 5 | 5
Weight decreased (Investigations) | 0 | 2 | 2 | 5
Amylase increased (Investigations) | 3 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 2 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram ambulatory abnormal (Investigations) | 0 | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
High density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 0
Blood calcitonin increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 1 | 0 | 0
Gastric pH decreased (Investigations) | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03353350/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03353350/SAP_001.pdf